CLINICAL TRIAL: NCT06437522
Title: A Phase II Clinical Trial To Evaluate the Efficacy and Safety of BL-B01D1+PD-1 Monoclonal Antibody in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (Non-nasopharyngeal Carcinoma) and Other Solid Tumors
Brief Title: A Study of BL-B01D1+PD-1 Monoclonal Antibody in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma and Other Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-204-02
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive BL-B01D1 + PD-1 monoclonal antibody as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1; Drug: PD-1 monoclonal antibody

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
Drug: PD-1 monoclonal antibody — Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This study is a phase II clinical study to explore the efficacy and safety of BL-B01D1 + PD-1 monoclonal antibody combination therapy in patients with recurrent or metastatic head and neck squamous cell carcinoma (non-nasopharyngeal carcinoma) and other solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subject volunteered to participate in the study and signed an informed consent;
2. Male or female aged ≥18 years and ≤75 years;
3. Expected survival time ≥3 months;
4. ECOG score 0-1;
5. Patients with recurrent or metastatic head and neck squamous cell carcinoma (non-nasopharyngeal carcinoma) and other solid tumors confirmed by histopathology and/or cytology;
6. Patients must provide a documented tumor tissue specimen of the primary or metastatic tumor within 3 years for PD-L1 testing and other testing;
7. At least one measurable lesion meeting the RECIST v1.1 definition was required;
8. No blood transfusion and no use of cell growth factors and/or platelet-raising drugs within 14 days before screening, and the organ function level must meet the requirements;
9. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
10. For premenopausal women of childbearing potential, a pregnancy test must be performed within 7 days before the initiation of treatment, a serum or urine pregnancy test must be negative, and the patient must not be lactating; All enrolled patients should take adequate barrier contraception during the entire treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Prior treatment with an ADC drug with TOP I inhibitors as a toxin;
2. Before the first delivery within four weeks or five half-life used anti-tumor treatment; Palliative radiotherapy was given within 2 weeks before the first dose;
3. Received any previous systemic antitumor regimen for solid tumors such as recurrent or metastatic head and neck squamous cell carcinoma;
4. Had received immunotherapy and developed ≥ grade 3 irAE or ≥ grade 2 immune-related myocarditis;
5. Use of an immunomodulatory drug within 14 days before the first dose of study drug;
6. Systemic corticosteroids were required within 2 weeks before the first dose of the study;
7. Has a history of severe disease of heart head blood-vessel;
8. Active autoimmune and inflammatory diseases;
9. Other malignant tumors that progressed or required treatment within 3 years before the first dose;
10. With ILD requiring steroid treatment, current ILD, or suspected ILD at screening;
11. Presence of: a) poorly controlled diabetes mellitus before study treatment; b) poorly controlled hypertension; c) history of hypertensive crisis or hypertensive encephalopathy;
12. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening;
13. Patients with active central nervous system metastasis;
14. Patients with pleural effusion, pericardial effusion or ascites with clinical symptoms or requiring repeated drainage;
15. Had allergic history to recombinant humanized antibody or human-mouse chimeric antibody or to any of BL-B01D1's excipients;
16. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
17. Human immunodeficiency virus antibody positive, active tuberculosis, active hepatitis B virus infection or active hepatitis C virus infection;
18. Active infection requiring systemic therapy;
19. Had participated in another clinical trial within 4 weeks before the first dose;
20. Who have a history of psychotropic drug abuse and cannot abstain from it or have mental disorders;
21. Other circumstances that the investigator deemed inappropriate for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-B01D1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BIRC is defined as the time between the date subjects are randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.

CONTACTS AND LOCATIONS:
Overall Officials: Chaosu Hu, Principal Investigator — Fudan University; Dongmei Ji, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China